CLINICAL TRIAL: NCT04240288
Title: Randomized Controlled Trial of Procalcitonin-Guided Antibiotic Therapy Versus Standard of Care for Complicated Intra-Abdominal Infections
Brief Title: Procalcitonin Guided Antibiotic Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAS5105
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Intra-Abdominal Infections
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Masking Description: Not applicable. The study is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other): Participants randomized to the control arm will be managed with the current standard of care including daily white blood cell count and vital sign documentation. The control group will also have daily procalcitonin levels drawn but the results will not be used to make decisions regarding antibiotic duration. Antibiotics will be given orally or intravenously at the discretion of the treating physician and will be given for a 10-day course, the current standard of care.
  Interventions: Other: Standard of Care Antibiotic Treatment
- Treatment Arm (Experimental): These participants will be managed with procalcitonin-guided antibiotic therapy. An index procalcitonin will be drawn within 24 hours of admission followed by daily procalcitonin levels. Per standard of care, patients will have daily white blood cell counts drawn and regular vital sign documentation. Antibiotics will be given orally or intravenously at the discretion of the treating physician. Antibiotics in this arm will be stopped once the procalcitonin value drops to ≤80% of its index value or to <0.5 ng/ml. Extension of antibiotics for more than 24 hours past this time will be documented.
  Interventions: Other: Procalcitonin-guided antibiotic treatment

INTERVENTIONS:
Other: Procalcitonin-guided antibiotic treatment — Antibiotics will be administered based on the procalcitonin lab results.
  Arms: Treatment Arm
Other: Standard of Care Antibiotic Treatment — Antibiotics will be administered based on standard of care treatment. The treating physicians will determine the treatment course.
  Arms: Control Arm

SUMMARY:
The overuse of antibiotics is an enormous problem facing the healthcare system both in the United States and across the world. The investigators plan to test the hypothesis that using procalcitonin levels (blood test) to guide the length of antibiotic therapy in patients with complicated intra-abdominal infections leads to shorter antibiotic treatment courses.

DETAILED DESCRIPTION:
A 2019 Centers for Disease Control (CDC) report describes the rate of antibiotic resistance as alarmingly high and says clinicians must make efforts to lower the development of resistance through more discerning antibiotic use. Complicated intra-abdominal infections (CIAIs), defined as an infection that extends beyond the hollow viscus of origin and into the peritoneal space, are a common problem with a 9.2% mortality rate worldwide, a morbidity of 5-50% and a 21.5% risk of extra-abdominal infections. The basic principles for treatment of CIAIs include source control and appropriate antibiotic coverage; however, source control cannot always be achieved in CIAIs, i.e. diverticular or appendiceal abscesses. The STOP-IT trial concluded that shorter courses of antibiotics for CIAIs with source control are equivalent to the traditional longer courses with regard to recurrent infections and mortality, even in the setting of sepsis, but the optimal duration of antibiotic treatment is unknown for patients with CIAIs without source control. Due to lack of guidelines, these patients are routinely treated with long antibiotic courses. Given the association of prolonged antibiotic courses and increased rates of post-treatment infectious complications and antimicrobial resistance, the Infectious Disease Society of America and the Surgical Infection Society acknowledge that there is an urgent need to study the appropriate duration of antimicrobial therapy for CIAIs. The biomarker procalcitonin is expressed by human epithelial cells in response to bacterial infections, distinguishes true bacterial infection from Systemic Inflammatory Response Syndrome (SIRS) and has been used in studies to identify CIAIs.

Procalcitonin-guided antibiotic management has been shown to decrease the number of antibiotic days in respiratory infections and reduce mortality among medical and surgical Intensive Care Unit (ICU) populations (including those with CIAIs). However, there is little data evaluating its role in guiding antibiotic therapy specifically for CIAIs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Ability to give consent in English or Spanish
* Imaging proven intra-abdominal infection (CT, US, and/or MRI)

Exclusion Criteria:

* Unable to give informed consent
* Patients enrolled in another trial
* Those having surgery for source control
* Patients with anastomotic leak
* Unable or unwilling to return or be contacted for clinical follow-up visits
* Currently incarcerated in a detention facility or in police custody
* Conditions with altered immune response or at risk for bacterial seeding
* Immunodeficiency (e.g., absolute neutrophil count <500/mm3, chronic immunosuppressive drugs, active chemotherapy or plans for chemotherapy in the following 30 days, or known AIDS [CD4 count <200 or AIDS-defining illness within the last year] assessed by patient history)
* Uncompensated liver failure
* Taking medication to treat active inflammatory bowel disease
* Malignancy, not in remission (ongoing chemotherapy patients excluded)
* Pregnant or expectation of becoming pregnant in the 30 days following baseline/screening
* Expected concurrent hemodialysis, peritoneal dialysis, or treatments using indwelling venous catheters
* Recent (within 90 days) placement of surgical implant (e.g., pacemaker, joint prosthesis, mechanical valve)
* Indwelling Left Ventricular Assist Device
* Patients with another infection (e.g., pneumonia, urinary tract infection) that requires treatment with another antibiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Number of Antibiotic Treatment Days | Up to 10 days
  The total number of antibiotic treatment days will be calculated for participants in both arms. Patients in the experimental arm will have their antibiotics stopped when the procalcitonin drops to ≤80% of its index value or to <0.5 ng/ml.

SECONDARY OUTCOMES:
Total Number of Recurrent Intra-Abdominal Infections or Extra-Abdominal Infections | Day 30
  To describe the rate of recurrent intra-abdominal infections in both the procalcitonin-guided antibiotic therapy arm and the control group. This will serve as a secondary outcome as well as a safety endpoint. We will describe the rate of antibiotic failure at 30 days, the 30-day mortality and the rate of extra-abdominal infections.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Fischkoff, MD, Principal Investigator — Columbia University